CLINICAL TRIAL: NCT00018733
Title: Biological Aspects of Depression and Antidepressant Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: MHBS-031-99F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Paroxetine; Desipramine

INTERVENTIONS:
Drug: paroxetine
Drug: Desipramine

SUMMARY:
This study will be measuring changes in depressive symptoms over a 7 week time period. Double-blind placebo controlled trial using the pharmacologic agents Paroxetine or Desipramine.

ELIGIBILITY:
* Diagnosis of major depressive disorder Ham-D Score > 18
* English speaking with ability to read and sign an informed consent

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1996-09; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Steve Brannan, M.D.; Cheryl Gonzalez, M.D.
Locations (1):
- South Texas Veterans Health Care System, San Antonio, Texas, United States